CLINICAL TRIAL: NCT06915142
Title: An Phase II Clinical Study on the Safety, Tolerability and Efficacy of HRS-7058 in Combination With Antitumor Drugs in Subjects With Solid Tumors
Brief Title: A Phase II Clinical Study of HRS-7058 in Combination With Antitumor Drugs in Patients With Advanced Malignant Tumour
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-7058-201
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-04

CONDITIONS: Advanced Malignant Tumour
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- HRS-7058 + SHR-1316 (Experimental)
  Interventions: Drug: HRS-7058 + SHR-1316
- HRS-7058 + SHR-1316 + Platinum-containing doublet chemotherapy (Experimental)
  Interventions: Drug: HRS-7058 + SHR-1316 + Platinum-containing doublet chemotherapy
- HRS-7058 + Cetuximab (Experimental)
  Interventions: Drug: HRS-7058 + Cetuximab
- HRS-7058 + SHR-1826 (Experimental)
  Interventions: Drug: HRS-7058 + SHR-1826
- HRS-7058 + SHR-1826 + SHR-1316 (Experimental)
  Interventions: Drug: HRS-7058 + SHR-1826 + SHR-1316
- HRS-7058 + SHR-A1202 (Experimental)
  Interventions: Drug: HRS-7058 + SHR-A1202
- HRS-7058 + BP102 (Experimental)
  Interventions: Drug: HRS-7058 + BP102
- HRS-7058 + SHR-9839 (Experimental)
  Interventions: Drug: HRS-7058 + SHR-9839
- HRS-7058 +SHR-A2102 +SHR-1316 (Experimental)
  Interventions: Drug: HRS-7058 +SHR-A2102 +SHR-1316
- HRS-7058 +SHR-9839(sc)+SHR-1316 (Experimental)
  Interventions: Drug: HRS-7058 +SHR-9839(sc)+SHR-1316
- HRS-7058 +SHR-1316 +BP102 (Experimental)
  Interventions: Drug: HRS-7058 +SHR-1316 +BP102
- HRS-7058 +SHR-A2102 +BP102 (Experimental)
  Interventions: Drug: HRS-7058 +SHR-A2102 +BP102
- HRS-7058 +SHR-A2102 +SHR-1316 +BP102 (Experimental)
  Interventions: Drug: HRS-7058 +SHR-A2102 +SHR-1316 +BP102

INTERVENTIONS:
Drug: HRS-7058 + SHR-1316 — HRS-7058 + SHR-1316
  Arms: HRS-7058 + SHR-1316
Drug: HRS-7058 + SHR-1316 + Platinum-containing doublet chemotherapy — HRS-7058 + SHR-1316 + Platinum-containing doublet chemotherapy
  Arms: HRS-7058 + SHR-1316 + Platinum-containing doublet chemotherapy
Drug: HRS-7058 + Cetuximab — HRS-7058 + Cetuximab
  Arms: HRS-7058 + Cetuximab
Drug: HRS-7058 + SHR-1826 — HRS-7058 + SHR-1826
  Arms: HRS-7058 + SHR-1826
Drug: HRS-7058 + SHR-1826 + SHR-1316 — HRS-7058 + SHR-1826 + SHR-1316
  Arms: HRS-7058 + SHR-1826 + SHR-1316
Drug: HRS-7058 + SHR-A1202 — HRS-7058 + SHR-A1202
  Arms: HRS-7058 + SHR-A1202
Drug: HRS-7058 + BP102 — HRS-7058 + BP102
  Arms: HRS-7058 + BP102
Drug: HRS-7058 + SHR-9839 — HRS-7058 + SHR-9839
  Arms: HRS-7058 + SHR-9839
Drug: HRS-7058 +SHR-A2102 +SHR-1316 — HRS-7058 +SHR-A2102 +SHR-1316
  Arms: HRS-7058 +SHR-A2102 +SHR-1316
Drug: HRS-7058 +SHR-9839(sc)+SHR-1316 — HRS-7058 +SHR-9839(sc)+SHR-1316
  Arms: HRS-7058 +SHR-9839(sc)+SHR-1316
Drug: HRS-7058 +SHR-1316 +BP102 — HRS-7058 +SHR-1316 +BP102
  Arms: HRS-7058 +SHR-1316 +BP102
Drug: HRS-7058 +SHR-A2102 +BP102 — HRS-7058 +SHR-A2102 +BP102
  Arms: HRS-7058 +SHR-A2102 +BP102
Drug: HRS-7058 +SHR-A2102 +SHR-1316 +BP102 — HRS-7058 +SHR-A2102 +SHR-1316 +BP102
  Arms: HRS-7058 +SHR-A2102 +SHR-1316 +BP102

SUMMARY:
This study is a multicentre, open phase II clinical study of dose escalation, dose extension and efficacy extension of HRS-7058 in combination with antitumor drugs in subjects with advanced malignant tumour. To evaluate the safety, tolerability and efficacy of HRS-7058 in combination with antitumor drugs.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects gave informed consent to the study before participating in, and voluntarily signed informed consent;
2. 18 to 75 years old (including both ends), gender is not limited;
3. Subjects with unresectable locally advanced or metastatic solid tumour confirmed by histopathology;
4. Having at least one evaluable or measurable lesion according to the solid tumour response Evaluation Criteria (RECIST 1.1);
5. ECOG Performance Status of 0 or 1;
6. The expected survival time is more than 12 weeks;
7. Be able to ingest drugs and be able to comply with trial and follow-up procedures;
8. Adequate bone marrow and organ function;
9. Female subjects of childbearing potential must undergo a serum pregnancy test within 7 days before the first administration of the study drug, and the result must be negative; and they must not be lactating. Female subjects of childbearing potential and male subjects whose partners are females of childbearing potential must agree to comply with contraceptive requirements from the time of signing the informed consent form until 5 months after the last administration of the study drug (for male subjects) or 8 months after the last administration of the study drug (for female subjects).

Exclusion Criteria:

1. Accompanied by untreated or active central nervous system (CNS) tumour metastasis;
2. Antitumor therapy within 28 days prior to initial use of the investigational drug;
3. The adverse reactions of previous anti-tumour therapy have not recovered to CTCAE ≤ grade 1;
4. With known or suspected interstitial pneumonia;
5. With severe cardiovascular and cerebrovascular disease
6. Had other malignancies within five years prior to first use of the investigational drug;
7. Severe infection within 28 days prior to first use of the investigational drug;
8. History of immune deficiency;
9. Refractory nausea, vomiting, or other gastrointestinal disorders that affect the use of oral medications;
10. The presence of uncontrolled pleural, abdominal or pericardial effusion;
11. Had undergone major organ surgery within 28 days prior to the first use of the study drug;
12. Women during pregnancy or lactation;
13. Known allergies and contraindications to the investigational drug or any of its components;
14. According to the judgment of the investigator, there are any other circumstances that may increase the risks of participating in the study, interfere with the study results, or make the subjects unsuitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) (Dose Escalation and Dose Expansion) | From the beginning of first patient in (FPI) to the end of dose expansion phase up to approximately 10 months
Safety endpoints: adverse events (AE) (Dose Escalation and Dose Expansion) | From the beginning of first patient in (FPI) to the end of dose expansion phase up to approximately 10 months]
Phase II recommended dose (RP2D)(Dose Escalation and Dose Expansion) | From the beginning of first patient in (FPI) to the end of dose expansion phase up to approximately 10 months]
Efficacy endpoints: Objective response rate (ORR) assessed based on RECIST v1.1 criterion (Efficacy Expansion) | From the beginning of first patient in (FPI) to the end of study up to approximately 32 months

SECONDARY OUTCOMES:
Efficacy endpoints: Objective response rate (ORR) assessed based on RECIST v1.1 criterion (Dose Escalation and Dose Expansion) | From the beginning of first patient in (FPI) to the end of dose expansion phase up to approximately 10 months
Efficacy endpoints: disease control rate (DCR) assessed based on RECIST v1.1 criterion (Dose Escalation and Dose Expansion) | From the beginning of first patient in (FPI) to the end of dose expansion phase up to approximately 10 months
Efficacy endpoints: duration of response (DoR) assessed based on RECIST v1.1 criterion (Dose Escalation and Dose Expansion) | From the beginning of first patient in (FPI) to the end of dose expansion phase up to approximately 10 months
Efficacy endpoints: progression-free survival (PFS) assessed based on RECIST v1.1 criterion (Dose Escalation and Dose Expansion) | From the beginning of first patient in (FPI) to the end of dose expansion phase up to approximately 10 months
Efficacy endpoints: overall survival (OS)(Dose Escalation and Dose Expansion) | From the beginning of first patient in (FPI) to the end of dose expansion phase up to approximately 10 months
Efficacy endpoints: disease control rate (DCR) assessed based on RECIST v1.1 criterion (Efficacy Expansion) | From the beginning of first patient in (FPI) to the end of study up to approximately 32 months
Efficacy endpoints: duration of response (DoR) assessed based on RECIST v1.1 criterion (Efficacy Expansion) | From the beginning of first patient in (FPI) to the end of study up to approximately 32 months
Efficacy endpoints: progression-free survival (PFS) assessed based on RECIST v1.1 criterion (Efficacy Expansion) | From the beginning of first patient in (FPI) to the end of study up to approximately 32 months
Efficacy endpoints: overall survival (OS) (Efficacy Expansion) | From the beginning of first patient in (FPI) to the end of study up to approximately 32 months
Safety endpoints: adverse events (AE)(Efficacy Expansion) | From the beginning of first patient in (FPI) to the end of study up to approximately 32 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided